CLINICAL TRIAL: NCT05429398
Title: A Single-arm, Open-label, Multicenter,Phase I Study of Linperlisib Combination With Camrelizumab in Patients With Advanced Solid Tumor
Brief Title: A Study of Linperlisib Combination With Camrelizumab in Patients With Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-013
Record Dates: First submitted 2022-05-05; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Advanced Solid Tumor
Keywords: PI3K inhibitor; PD-1 inhibitor; advanced solid tumor
MeSH Terms: interventions — camrelizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linperlisib +Camrelizumab 200mgQ3w (Experimental): Linperlisib will be administrated orally from 40mgQD, 60mgQD to 80mgQD in sequence during dose excalation part and a selected dose in dose expansion part,for 21 consecutive days as a treatment cycle; Camrelizumab will be administrated intravenously 200mg every 3 weeks in all patients just before the administration of Linperlisib.
  Interventions: Drug: Linperlisib Tablet

INTERVENTIONS:
Drug: Linperlisib Tablet — 1. Linperlisib Tablet Oral administration, once a day, for 21 consecutive days as a treatment cycle;
  2. Camrelizumab for Injection 200 mg intravenously every 3 weeks. Camrelizumab should be administered prior to Linperlisib.
  Other Names: Camrelizumab for Injection

SUMMARY:
It is a single-arm, open-label, multicenter, phase I trial,aiming at exploring the MTD and RP2D of Linperlisib combination with Camrelizumab in treating patients with advanced solid tumor,observing the preliminary efficacy.

DETAILED DESCRIPTION:
The trial can be divided into two parts: dose escalation part and dose expansion part.

Camrelizumab will be administrated intravenously in a predetermined fixed dose(200mgQ3w）in both parts.

In dose escalation part,Linperlisib will be administrated from 40mgQD,60mgQD to 80 mgQD in sequence with the classic "3+3" design.The purposes of this part are figuring out the MTD and RP2D of Linperlisib combination with Camrelizumab in treating patients with advanced solid tumor,and observing the PK characteristics of Linperlisib when using combination with Camrelizumab.

When finishing the dose escalation part,one combination dose of Linperlisib with Carelizumab will be selected to be studied on a wider scale of patients with advantage solid tumor in dose expansion part.Purposes of this part are further observing the PK characteristics of Linperlisib when using combination with Camrelizumab,while observing the preliminary efficacy of Linperlisib when using combination with Camrelizumab.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old≦age≦75 years old;
* Histologically or cytologically confirmed locally advanced or metastatic malignant solid tumors；
* Failure of previous standard treatment (sufficient prior treatment and no better treatment than participating in clinical research);
* Qualified basic organ function and body condition;
* The expected survival is greater than 3 months;
* Adequate washout period.

Exclusion Criteria:

* Prior allergy to study drug components;
* Chronic metabolic diseases that are poorly controlled by medication;
* Brain metastases, infection, hemorrhage, autoimmune disease or cardiovascular disease, whichever is in active state;
* Digestive tract diseases that affect absorption of studied drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
DLTs | At the end of Cycle 1 (each cycle is 21 days)
  dose limited toxicities
TEAEs | from day 1after taking the investigational product till 30 days after withdrew from the study
  treatment emergent adverse events

SECONDARY OUTCOMES:
Drug exposure | At the end of Cycle 1 (each cycle is 21 days)
  Peak Plasma Concentration (Cmax)
PK parameters | At the end of Cycle 1 (each cycle is 21 days)
  Area under the plasma concentration versus time curve (AUC).etc.
Effectiveness evaluation index | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  ORR、DOR、DCR、TTR、PFS、OS

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Cancer Hospital affiliated to Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No